CLINICAL TRIAL: NCT04050904
Title: Chronic Heart Failure Therapy Optimization With CardioRenal Remote Monitoring System (HERMESHF)
Acronym: HERMESHF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CardioRenal (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CR-2018-001
Record Dates: First submitted 2019-05-17; First posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Heart Failure
Keywords: heart failure; algorithm
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Prospective single-arm open pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ExpHeart (Experimental): The Information System is a cyber-securised web application and the Expert System uses a proprietary therapeutic algorithm to optimize pharmacological HF treatment.
  Interventions: Device: ExpHeart

INTERVENTIONS:
Device: ExpHeart — ExpHeart is composed of an Information System (web application) and an algorithm, the Expert System, embedded on the Information System. The Information System is a cyber-securised web application and the Expert System uses a proprietary therapeutic algorithm to optimize pharmacological HF treatment. The Expert System is based on the analysis of a continuously updated clinical database integrating the patient's electronic medical record (managed by the Information System). The Expert System will generate prescription recommendations directed to the treating investigator through the Information System.

SUMMARY:
This clinical study evaluates short-term feasibility and safety of CardioRenal ExpHeart in patients with worsening heart failure with reduced ejection fraction to optimize pharmacological heart failure treatment.

DETAILED DESCRIPTION:
The study will take place as follows :

The remote monitoring of the biomarkers (5 days a week, between 7am - 12 midday). The home-based monitoring of congestion by Hb and Hte, eGFR using the CKD EPI formula (creatinine) and potassium variables will be measured with point of care devices, after minimally invasive blood sampling operated by the healthcare professional who will manually enter the data in the Information System.

2. ExpHeart is composed of an Information System (web application) and an algorithm, the Expert System, embedded on the information system. The Information System is a cyber-securised web application and the Expert System uses a proprietary therapeutic algorithm to optimize pharmacological HF treatment. The Expert System is based on the analysis of a continuously updated clinical database integrating the patient's electronic medical record (managed by the Information System). The Expert System will generate prescription recommendations directed to the treating investigator through the Information System. The Expert System recommendations are based on ESC clinical guidelines (Annex II). This evaluated solution Expheart is not CE marked yet.

3. Decision on treatment update and/or optimization will be operated by physicians and healthcare professionals who will monitor compliance with the study protocol including the smooth functioning of bilateral patientinvestigator communication, i.e. (i) receipt by the investigator of recommendations from Expheart solution, (ii) adequate action/decision of the investigator and (iii) implementation of the appropriate action at the patient level.

The Investigator will inform the patient's treating physician/General practitioner (by phone and mail) about the participation of his/her patient to the study and will inform him that any HF treatment prescription change will be performed by him/her during the study period.

Moreover, in case of any technical difficulty, assistance will be provided by a dedicated call center, serviced daily by the promotor (Monday to Friday, support@cardio-renal.com).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who understand the study procedures and agree to participate by providing informed consent.
* Male or female aged ≥18 years
* Subjects with worsening HF:

  1. Currently admitted to hospital with worsening heart failure, OR
  2. Discharged within 2 weeks from hospitalization with worsening heart failure AND
  3. HF with reduced ejection fraction (i.e. ejection fraction ≤ 35% documented within 6 months before enrolment)
  4. NT-proBNP > 1000 pg/ml, or BNP > 200 pg/ml. For subjects with atrial fibrillation, BNP must be > 700 pg/ml or NT-proBNP > 2500 pg/ml.
  5. Receiving suboptimal therapy i.e. no doses or doses < 50% of guideline target optimal of ACE inhibitors or ARB or ARNI or MRA (as per ESC guidelines recommendations, Annex II) AND at risk of developing hyperkalaemia or worsening renal function i.e. ANY of the following:

     1. documented history of hyperkalaemia or of worsening renal function leading to ACE-I or ARB or ARNI or MRA down-titration or discontinuation,
     2. age > 75 years,
     3. eGFR < 50 ml/min/1.73 m2 anytime during hospitalization (using the CKD EPI formula),
     4. diabetes.

Exclusion Criteria:

* Subjects with newly diagnosed heart failure within the past 3 months.
* Subjects known to be poorly adherent to their HF medications/treatment regimen.
* Subjects who have had a non-cardiac surgical procedure or cardiac-related interventional procedure (for example but not limited to angiogram, CABG, angioplasty or pacemaker insertion) within the past 30 days.
* Subjects who have had an ACS, or MI, within the past 30 days.
* Subjects with eGFR <30 ml/min/1.73m2 (using CKD EPI formula)
* Subjects with life expectancy less than 3 months in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08-15 (Estimated); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Hospitalization | 5 weeks
  All cause hospitalization (total number of participants hospitalized for any cause)
Mortality (number of all cause death) | 5 weeks
  All cause death
Heart failure hospitalization (number of patients hospitalized for heart failure) | 5 weeks
  Heart failure hospitalization defined as:
  * Heart failure related visit to an emergency room
  * Heart failure related visit to an ambulatory heart failure care
  * Heart failure related hospital admissions
Hyperkalemia (number of participants with episode of hyperkaliemia) | 5 weeks
  Hyperkalemia >6 mmol/L (confirmed by immediate recheck on site with vein puncture by the study nurse)
Hypokalemia (number of participants with episode of hypokaliemia) | 5 weeks
  Hypokalemia <3.5 mmol/L (confirmed by immediate recheck on site with vein puncture by the study nurse)
Renal function | 5 weeks
  Number of participants with at least one episode of worsening renal function >50 %, >100 %
Feasibility outcome | 5 weeks
  Number of successful procedures during each study steps from puncture and sampling process to implementation of the specific action at the patient level

OTHER OUTCOMES:
Pharmacotherapy | 5 weeks
  Number of participants with changes from baseline to 5 weeks post enrollment of doses of ACE inhibitors or ARB or ARNI or MRAs and of loop diuretics
Dose titration | 5 weeks
  Frequency of dose titration of ACE inhibitors or ARB or ARNI or MRAs and of loop diuretics
Rate of patients with optimal therapy | 5 weeks
  Rate of patients receiving optimal therapy of ACE inhibitors or ARB or ARNI or MRAs (i.e. receiving doses > 50% of guideline target doses), alive, and not hospitalized for heart failure
Congestion | 5 weeks
  Changes from baseline to 5 weeks post enrollment in congestion score as assessed by lung comet ultrasound
Changes in BNP | 5 weeks
  Changes from baseline to 5 weeks post enrollment in blood levels of BNP (pg/mL)
Hemoglobin | 5 weeks
  Changes from baseline to 5 weeks in blood hemoglobin concentration (g/L)
Hemoglobin | 5 weeks
  Changes from baseline to 5 weeks in hematocrit (%)
Renal function | 5 weeks
  Changes from baseline to 5 weeks in eGFR (ml/min/1.7 m2) (using the CKD EPI formula)
Blood potassium | 5 weeks
  Changes from baseline to 5 weeks in blood potassium (mmol/L)
Patient experience | 5 weeks
  Sociology survey with questionnaire on subjective experience (Optional sub-study) Changes from baseline to 5 weeks in Health-related Quality of life, measured using the Kansas City Cardiomyopathy Questionnaire (KCCQ)
Exploratory pathophysiological outcomes | 5 weeks
  Correlation between changes in Hb and hematocrit with the following parameters:
  * BNP changes from baseline (pg/mL)
  * Lung comet changes (congestion score as assessed by lung comet ultrasound)
  * HF-related visit to an emergency room (number of visits)
  * HF-related visit to an ambulatory HF care unit (number of visits)
  * HF-related hospital admissions (number of days of hospitalizations)
  * HF-related death (number of deaths due to HF)
  * Administration of an intravenous diuretic (dose of intravenous diuretic)
  * Increase in dose of, or addition of a new, oral diuretic

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Mebazaa, MD, Principal Investigator — Hôpital Lariboisière

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Official Website of CardioRenal — https://www.cardio-renal.com/